CLINICAL TRIAL: NCT05993858
Title: A Single-Center, Single-Arm Exploratory Clinical Trial of Neoadjuvant PD-1 Inhibitor Combined With Cetuximab in Operable Locally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: Neoadjuvant PD-1 Inhibitor Combined With Cetuximab in Operable Locally Advanced HNSCC
Acronym: PC-1
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UHCT230527
Record Dates: First submitted 2023-07-19; First posted 2023-08-15 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-07

CONDITIONS: Head and Neck Squamous Cell Carcinoma; Neoadjuvant Therapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — toripalimab; Cetuximab; Surgical Procedures, Operative; Radiotherapy; Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant therapy+Surgery+Adjuvant therapy+Consolidation therapy (Other): Participants receive totally 3 cycles of neoadjuvant therapy (Toripalimab+cetuximab), then radical treatment(surgery). After surgery, Participants receive radiotherapy or chemoradiotherapy according to the pathological results of the operation. Then, participants receive consolidation therapy of Toripalimab.
  Interventions: Drug: 3cycles (Toripalimab + cetuximab); Procedure: Surgery; Radiation: Radiotherapy or chemoradiotherapy

INTERVENTIONS:
Drug: 3cycles (Toripalimab + cetuximab) — Toripalimab by intravenous (IV) infusion every 3 weeks (Q3W), 3 preoperative and 17 consolidated doses.
  The preoperative starting dose of cetuximab is 400 mg/m^2 by IV infusion over 120 minutes for 1 week, subsequently followed by 250 mg/m^2 IV infusion over 60 minutes, from week 2 to 9.
Procedure: Surgery — After neoadjuvant therapy, patients would accept surgery within 11-13 weeks.
Radiation: Radiotherapy or chemoradiotherapy — Adjuvant radiotherapy was given 4 weeks after surgery. Patients with positive intraoperative pathological margins/extra lymph node envelope invasion are treated with an additional cisplatin synchronous chemotherapy.

SUMMARY:
This is a single-center, single-arm, phase II clinical study to evaluate the efficacy and safety of PD-1 inhibitor combined with cetuximab in neoadjuvant therapy for locally advanced HNSCC.

DETAILED DESCRIPTION:
At present, the standard treatment for patients with operable locally advanced head and neck squamous cell carcinoma (HNSCC) is adjuvant radiotherapy with or without platinum-based synchronous chemotherapy after operation. However, the risk of recurrence, metastasis and death remains high in this population with this intense combination treatment regimen. Both EGFR monoclonal antibody and PD-1 inhibitors have proven the effect in advanced HNSCC. At the same time, cetuximab and PD-1 inhibitors have been reported to have a synergistic effect that may improve patient survival. This study aims to explore the efficacy and safety of PD-1 inhibitor combined with cetuximab in neoadjuvant therapy for locally advanced HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* The age at the time of enrollment is more than 18 years old and less than 70 years old, both male and female.
* Histologically diagnosed as squamous cell carcinoma of the mouth, oropharynx, hypopharynx or larynx; preoperative evaluation can be surgically resected.
* Have the following high-risk recurrence conditions as defined in the 8th edition of the American Joint Committee on Cancer [AJCC] Guidelines: a)HPV-negative disease, stage III, IVa, according to the head and Neck Tumor/lymph node/metastasis (TNM) guidelines; b)non-oropharyngeal HPV-positive disease, stages III, IVa, IVb, according to head and neck TNM guidelines.
* No previous treatment for HNSCC.
* Have at least one evaluable target lesion according to RECIST version 1.1 criteria.
* The Eastern Cancer Cooperation Organization (ECOG) physical fitness score was 0 or 1.
* Major organs have normal function, the following criteria are met:
* The standard of blood routine examination（(not transfused or receiving component blood within 14 days prior to testing)：hemoglobin (HB) ≥ 9g/dL；absolute neutrophil count (ANC) ≥1.5×10^9/L, platelets (PLT) ≥100×10^9/L.
* Biochemical examination: serum total bilirubin (TBIL) <1.5 times the upper limit of normal value(ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT)<2.5 ULN; serum creatinine≤ULN and endogenous creatinine clearance>50 mL/min (Cockcroft-Gault formula) Gault formula).
* Signed written informed consent.
* Adhere to the research protocol judged by the investigator.
* female subjects of reproductive potential must have a negative serum pregnancy test prior to the first dose of the trial drug.
* The male fertile patients and female fertile patients with pregnancy risk must consent to the use of 2 contraceptive methods (at least one of which is considered highly effective) throughout the study period.
* Patients who are willing and able to follow visit schedules, treatment plans, laboratory tests, and other research procedures.

Exclusion Criteria:

* prior treatment with EGFR/PD-1/PD-L1/PD-L2/CD137/CTLA-4 antibodies(including ipilimumab) or activating or inhibitory agents targeting T-cell receptors.
* Major surgery within 4 weeks before enrollment.
* Proven allergic to EGFR monoclonal antibody, PD-1 antibody or its excipients.
* Any active autoimmune disease or history of autoimmune disease (e.g., the following: interstitial pneumonia, uveitis, enteritis, hepatitis, hypophysitis, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism (can be included after effective hormone replacement therapy), etc; patients with vitiligo or asthma in complete remission in childhood may be included, adults patients with asthma who do not need any intervention and require medical intervention with bronchodilators may be included) .
* Previous or co-existing malignancies (except those that have been cured and have survived cancer-free for more than 5 years, such as basal cell carcinoma of the skin, carcinoma in situ of the cervix, and papillary carcinoma of the thyroid).
* Failure to control cardiac clinical symptoms or disease, e.g., the following: a) patients with NYHAII or above heart failure, b) unstable angina pectoris c) patients with myocardial infarction within 1 year, d) patients with clinically significant supraventricular or ventricular arrhythmias requiring clinical intervention.
* Subjects requiring systemic treatment with corticosteroids (> 10mg/ day prednisone efficacy dose) or other immunosuppressants within 14 days prior to administration of the study drug were allowed to use inhaled or topical steroids and adrenal hormone replacement at a dose>10mg/day prednisone efficacy dose in the absence of active autoimmune disease.
* Have active infections that require treatment.
* Have a congenital or acquired immune deficiency (such as HIV infection), active hepatitis B (HBV-DNA≥10^3 copy number/ml), or hepatitis C (hepatitis C antibody positive and HCV-RNA above the lower detection limit of analytical methods).
* The patient has received other treatment before.
* Had received live vaccine within 4 weeks prior to starting study treatment.
* A known history of psychotropic substance abuse, alcohol or drug use.
* Pregnant or lactating women.
* In the investigator's judgment, the subjects had other factors that might have led to their forced discontinuation of the study, such as other serious medical conditions (including mental illness) requiring concomitant treatment, serious abnormalities in laboratory test values, or family or social factors that might have affected the safety of the subjects or the circumstances of the trial data collection.
* HNSCC Patients with T1/T2 or N0/N1.
* oral cancer, larynx cancer, hypopharyngeal cancer withT4b or N3 and P16-oropharyngeal cancer.
* Have active pulmonary tuberculosis.
* Serious infections (including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia) that occurred within 4 weeks prior to initiation of study treatment.
* Had received systemic immunostimulatory drugs (including but not limited to interferon or interleukin-2 [IL-2]) within 4 weeks prior to initiation of study therapy or remained within 5 drug half-lives (choice the longer of the two).
* Patients with recurrent peptic ulcers (e.g., gastric ulcers, duodenal ulcers), who have a history of peptic ulcer complications such as perforation, bleeding, obstruction, etc., or who have been assessed by clinicians as having a higher risk of complications.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-10-20 (Estimated); Primary Completion 2025-12-20 (Estimated); Study Completion 2026-12-20 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) Rate evaluated by investigators | up to 13 weeks after neoadjuvant
  pCR rate is defined as the percentage of participants having an absence of residual invasive cancer in resected tumour and lymph nodes following completion of neoadjuvant therapy.

SECONDARY OUTCOMES:
2 years Event-free survival (EFS) Rate evaluated by investigators | EFS Up to 3 years
  Event Free Survival (EFS): EFS is defined as the time from randomization until radiographic disease progression, local progression precluding surgery, inability to resect the tumor, local or distant recurrence, or death due to any cause. The 2y-EFS rate is defined as the probability of event-free survival for a patient at a given point in time (2 years).
Incidence of AEs/SAEs | Up to 3 years
  Overall incidence of adverse events (AEs); incidence of grade 3 and above AEs; incidence of serious adverse events (SAEs).
Objective Response Rate (ORR) evaluated by investigators | Up to 3 years
  The ORR was defined as proportion of patients whose tumor volume was reduced to 30% and sustained for more than 4 weeks as assessed by RECIST 1.1.
Major Pathological Response (MPR) Rate evaluated by investigators | up to 13 weeks after neoadjuvant
  MPR rate is defined as the percentage of participants having ≤10% viable tumor cells in the resected primary tumor and all resected lymph nodes in neoadjuvant therapy.
2 years Disease-free survival (DFS) Rate evaluated by investigators | DFS Up to 3 years
  DFS is defined as the time from postoperation until radiographic disease progression, local or distant recurrence, or death due to any cause. The 2y-DFS rate is defined as the probability of disease-free survival for a patient at a given point in time (2 years).
Organ Retention Rate | Up to 3 years
  Organ retention rate is defined as the proportion of patients whose tumor avoids radical surgery.

OTHER OUTCOMES:
Exploratory analysis of the tumor microenvironment related with the outcome | Up to 3 years
  Exploratory analysis of the tumor microenvironment related to the outcome(including the number, function and metabolism of immune cells in tumor microenvironment).
Exploratory analysis of potential biomakers related with the outcome | Up to 3 years
  Exploratory analysis of potential biomarkers related to the outcome (including PD-L1 expression in tissue specimen, tumor mutation burden (TMB), whole exome sequencing (WES) ,Single-cell RNA-sequencing (scRNA-seq) and Spatial transcriptomics (ST)).

CONTACTS AND LOCATIONS:
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hebei, China